CLINICAL TRIAL: NCT06833840
Title: Evaluation of the Prognostic Role of SOX2 as a Tumor Stem Cell Marker in Odontogenic Cysts and Tumors
Brief Title: Evaluation of the Expression and Prognostic Role of Tumor Stem Cell Marker SOX2 in Odontogenic Cysts and Tumors
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: A06010222
Record Dates: First submitted 2025-01-21; First posted 2025-02-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Odontogenic Cysts; Odontogenic Tumors
Keywords: Ameloblastoma; odontogenic keratocyst; dentigerous cyst; SOX2; immunohistochemistry
MeSH Terms: conditions — Odontogenic Cysts; Odontogenic Tumors; Ameloblastoma; Dentigerous Cyst

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ameloblastoma group: patients diagnosed with ameloblastoma
- Odontogenic keratocyst group: patients diagnosed with Odontogenic keratocyst
- Dentigerous cyst group: patients diagnosed with Dentigerous cyst

SUMMARY:
The pathogenesis of odontogenic lesions remains unclear; however, a probable explanation may involve the existence of tumor stem cells (TSCs), which are thought to generate both benign and malignant tumors. The preservation of stem cells during early dental development is governed by many transcription factors, including sex-determining region Y (SRY)-box 2 (SOX-2). Numerous studies observed the increased expression of SOX2 in various benign and malignant tumors, as its impact on tumorigenesis varies according to tumor type. The purpose of this study is to assess the immunoexpression of the stem cell marker SOX2 in diverse types of odontogenic cysts and tumors in order to identify its prognostic significance and to show if it correlates to clinicopathologic parameters of those odontogenic lesions.

DETAILED DESCRIPTION:
Forty-five surgical specimens were included in this study: 15 ameloblastomas (Ab), 15 odontogenic keratocysts (OKC), and 15 dentigerous cysts (DC). An immunohistochemical (IHC) study using the SOX2 Rabbit Polyclonal Antibody was done, and SOX2 expression was evaluated by two methods: computer-assisted digital image analysis to measure staining surface area percentage and a semi-quantitative method for subjectively scoring percentage and intensity of SOX2 staining. Positive specimens were considered when the nucleus had brown staining.

ELIGIBILITY:
Inclusion criteria:

1. Patients with benign odontogenic cysts and tumors which presented either in Maxilla or Mandible ( as indicated by incisional biopsies )

Exclusion criteria:

1. Patients with systemic diseases that absolutely contraindicate surgical procedures.
2. Malignant odontogenic tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male and female
Study Population: Patients in the Outpatient Clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
SOX2 staining score | 6 months
  Semi-quantitative method for subjectively scoring the immunohistochemical staining. Positive specimens were considered when the nucleus had brown staining.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No